CLINICAL TRIAL: NCT01622231
Title: Study FFR116365, an Open-label Study of GW685698X in Paediatric Subjects With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116365
Record Dates: First submitted 2012-06-07; First posted 2012-06-19 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — fluticasone furoate

ARMS (1):
- GW685698X (Experimental): GW685698X 55mcg/day
  Interventions: Drug: Fluticasone furoate

INTERVENTIONS:
Drug: Fluticasone furoate — 55 mcg/day, intranasal, 12 weeks

SUMMARY:
Safety of GW685698X (55 µg/day, q.d.) nasal spray over a period of 12 weeks in Japanese paediatric subjects ages 2 to < 15 years with perennial allergic rhinitis will be evaluated. And secondarily, efficacy and systemic exposure of GW685698X (55 µg/day, q.d.) nasal spray over a period of 12 weeks in Japanese paediatric subjects ages 2 to < 15 years with perennial allergic rhinitis will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* 2 to <15 years of age, male or eligible female (females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control), outpatient
* Diagnosis of perennial allergic rhinitis: A positive test response to house dust and/or dust mites on serum antigen-specific IgE antibody test at Visit 1. Six months or more clinical history of perennial allergic rhinitis. A positive test result on nasal eosinophil count at Visit 1/1A.
* Either subject's parent/guardian who signed ICF or subject is able to complete assessments on the patient diary through the study.
* ALT < 2xULN; alkaline phosphatase and bilirubin <= 1.5xULN
* Average of 3TNSS is >= 3.0 in the last consecutive 4 days prior to Visit 2.
* Completion of the patient diary on >= 3 days of the last consecutive 4 days prior to Visit 2

Exclusion Criteria:

* Has a seasonal pollen as an allergen
* A nose disorder that could affect the assessment of the study medication or eye or nose surgery (within 3 months prior to Visit 1)
* Bacterial or viral infection of upper respiratory tract or eye
* Concurrent disease/abnormalities: Clinically significant uncontrolled disease
* Known hypersensitivity to corticosteroids or any excipients in the investigational product
* Has recent participation in a study and/or exposure to an investigational study drug within 3 months prior to Visit 1
* Use of the following medication and/or its combination drug within the specified time:

Anti-IgE (Within 6 months prior to Visit 1), Immunosuppressive medications or Systemic corticosteroids (Within 8 weeks prior to Visit 1), Topical corticosteroids (Within 4 weeks prior to Visit 1), Immunotherapy or nonspecific allassotherapy which was initiated, discontinued or changed its dose within 4 weeks prior to Visit 1

* Affiliation with Investigator's Site: Relative or employee
* History of alcohol or drug abuse, children in care or in the opinion of the investigator (sub-investigator), inappropriate to be enrolled in the study.
* Bacterial or viral infection of upper respiratory tract or eye during the screening period.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116365 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met the inclusion criteria at Visit 1/1A entered a Screening Period (Visit 1 to 2). Participants who met the eligibility criteria for randomization entered the Treatment Period (Visit 2 to 5), during which they received GW685698X 55 micrograms (µg) once daily (QD) for a period of 12 weeks.
Groups:
- GW685698X 55 μg QD: Participants received GW685698X nasal spray (55 micrograms [µg]) as one spray into each nostril (27.5 μg per spray) once daily (QD) in the morning for 12 weeks.
Period: Overall Study
Arm/Group | GW685698X 55 μg QD
Started | 61
Completed | 59
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (3.59)
Gender [Count of Participants; unit: Participants]
  Female | 19
  Male | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Non-serious Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an other important medical event, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs (occurring at a frequency threshold >=5%) and SAEs.
Time Frame: From the start of study treatment (Visit 2) until follow-up contact (Visit 6) (up to 13 weeks)
Population: Safety Population: all participants who received at least one dose of medication
Measure: Number; unit: participants
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
participants
  Any AE | 41
  Any SAE | 0

2. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophil Count at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline. Basophils, eosinophils, lymphocytes, monocytes, and total neutrophil counts are measured as the percentage of cells in white blood cells.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Percentage of cells
  Basophils, Week 4, n=60 | -0.08 (0.353)
  Basophils, Week 12/early withdrawal, n=61 | -0.12 (0.356)
  Eosinophils, Week 4, n=60 | -0.29 (2.538)
  Eosinophils, Week 12/early withdrawal, n=61 | -1.38 (2.991)
  Lymphocytes, Week 4, n=60 | -1.22 (6.863)
  Lymphocytes, Week 12/early withdrawal, n=61 | -1.77 (8.181)
  Monocytes, Week 4, n=60 | 0.24 (1.604)
  Monocytes, Week 12/early withdrawal, n=61 | 0.26 (1.714)
  Total Neutrophils, Week 4, n=60 | 1.36 (8.355)
  Total Neutrophils, Week 12/early withdrawal, n=61 | 3.02 (9.684)

3. Secondary Outcome: Change From Baseline in Hemoglobin at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Grams per liter (grams/L)
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Grams per liter (grams/L)
  Hemoglobin, Week 4, n=60 | -1.9 (7.34)
  Hemoglobin, Week 12/early withdrawal, n=61 | 0.1 (6.09)

4. Secondary Outcome: Change From Baseline in Platelet Count and White Blood Cell (WBC) Count at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: giga (10^9) cells (GI)/L
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
giga (10^9) cells (GI)/L
  Platelet count, Week 4, n=60 | -0.4 (54.95)
  Platelet count, Week 12/early withdrawal, n=61 | -2.9 (56.26)
  WBC count, Week 4, n=60 | -0.45 (1.860)
  WBC count, Week 12/early withdrawal, n=61 | -0.00 (2.092)

5. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: tera (10^12) cells (TI)/L
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
tera (10^12) cells (TI)/L
  RBC count, Week 4, n=60 | -0.081 (0.2386)
  RBC count, Week 12/early withdrawal, n=61 | -0.039 (0.2080)

6. Secondary Outcome: Change From Baseline in Hematocrit at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Proportion of RBCs in blood
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Proportion of RBCs in blood
  Hematocrit, Week 4, n=60 | -0.0061 (0.01965)
  Hematocrit, Week 12/early withdrawal, n=61 | -0.0062 (0.01824)

7. Secondary Outcome: Change From Baseline in Albumin and Total Protein at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: grams/L
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
grams/L
  Albumin, Week 4, n=60 | -1.4 (2.05)
  Albumin, Week 12/early withdrawal, n=61 | -0.8 (1.93)
  Total protein, Week 4, n=60 | -1.8 (3.41)
  Total protein, Week 12/early withdrawal, n=61 | -0.9 (3.36)

8. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Gamma Glutamyltransferase (GGT) at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: International units (IU)/L
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
International units (IU)/L
  ALP, Week 4, n=60 | -49.9 (89.43)
  ALP, Week 12/early withdrawal, n=61 | 88.5 (586.10)
  ALT, Week 4, n=60 | 0.7 (4.19)
  ALT, Week 12/early withdrawal, n=61 | 0.4 (4.72)
  AST, Week 4, n=60 | -0.3 (3.45)
  AST, Week 12/early withdrawal, n=61 | 0.2 (3.39)
  GGT, Week 4, n=60 | -0.1 (1.63)
  GGT, Week 12/early withdrawal, n=61 | 0.1 (1.95)

9. Secondary Outcome: Change From Baseline in Direct Bilirubin, Total Bilirubin, and Creatinine at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Micromoles (μmol)/L
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Micromoles (μmol)/L
  Direct bilirubin, Week 4, n=60 | 0.114 (0.9889)
  Direct bilirubin, Week 12/early withdrawal, n=61 | -0.028 (0.8545)
  Total bilirubin, Week 4, n=60 | 0.370 (2.2504)
  Total bilirubin, Week 12/early withdrawal, n=61 | -0.533 (2.2844)
  Creatinine, Week 4, n=60 | -1.6649 (5.21356)
  Creatinine, Week 12/early withdrawal, n=61 | -0.5797 (5.63473)

10. Secondary Outcome: Change From Baseline in Calcium, Chloride, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) at Week 4 and Week 12/Early Withdrawal
Description: Change from Baseline was calculated as the value at the post-Baseline time points minus the value at Baseline.
Time Frame: Baseline, Week 4, and Week 12/Early Withdrawal
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Millimoles (mmol)/L
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Millimoles (mmol)/L
  Calcium, Week 4, n=60 | -0.0541 (0.09085)
  Calcium, Week 12/early withdrawal, n=61 | -0.0372 (0.07480)
  Chloride, Week 4, n=60 | 1.3 (2.27)
  Chloride, Week 12/early withdrawal, n=61 | 1.1 (2.04)
  Potassium, Week 4, n=60 | -0.13 (0.378)
  Potassium, Week 12/early withdrawal, n=61 | -0.06 (0.380)
  Sodium, Week 4, n=60 | -0.4 (1.70)
  Sodium, Week 12/early withdrawal, n=61 | -1.2 (1.58)
  Urea/BUN, Week 4, n=60 | -0.4998 (1.12504)
  Urea/BUN, Week 12/early withdrawal, n=61 | -0.0954 (1.18765)

11. Secondary Outcome: Mean Change From Baseline in the 3 Total Nasal Symptom Score (3TNSS) Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the informed consent form (ICF) or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For the entire assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the mean score for the entire treatment period minus the score at Baseline.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Entire Treatment Period, n=61 | -2.2 (1.65)
  Week 1 to 2, n=61 | -1.6 (1.58)
  Week 3 to 4, n=61 | -2.5 (1.84)
  Week 7 to 8, n=60 | -2.4 (1.86)
  Week 11 to 12, n=60 | -2.0 (2.07)

12. Secondary Outcome: Mean Percent Change From Baseline in the 3 Total Nasal Symptom Score (3TNSS) Over the Entire Treatment Period, Week 1to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the informed consent form (ICF) or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For the entire assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from Baseline=(mean score at the post-Baseline assessment minus the score at Baseline) divided by the Baseline value * 100.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Percent change
  Entire Treatment Period, n=61 | -46.9 (33.25)
  Week 1 to 2, n=61 | -31.6 (36.36)
  Week 3 to 4, n=61 | -53.2 (36.81)
  Week 7 to 8, n=60 | -50.9 (38.00)
  Week 11 to 12, n=60 | -40.7 (41.58)

13. Secondary Outcome: Mean Change From Baseline (BL) in Daily Variation of the 3 Total Nasal Symptom Score (3TNSS)
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the informed consent form (ICF) or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The BL value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For the entire assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from BL was calculated as the mean score for the entire treatment period minus the score at BL. Only those participants available at the indicated time points were assessed.
Time Frame: Baseline, Day 1 to Day 84
Population: Full Analysis Set (FAS) Population: all participants meeting the primary criteria for enrollment, without any major good clinical practice (GCP) deviation, who received at least one dose of the assigned treatment and had diary assessment for 3TNSS after receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Day 1, n=61 | -0.5 (1.81)
  Day 2, n=61 | -0.8 (1.90)
  Day 3, n=61 | -0.9 (1.64)
  Day 4, n=61 | -1.3 (1.76)
  Day 5, n=61 | -1.4 (1.75)
  Day 6, n=61 | -1.3 (1.76)
  Day 7, n=61 | -1.6 (1.83)
  Day 8, n=61 | -1.9 (1.94)
  Day 9, n=61 | -1.9 (2.12)
  Day 10, n=61 | -2.0 (1.90)
  Day 11, n=61 | -1.8 (2.18)
  Day 12, n=61 | -1.9 (1.98)
  Day 13, n=61 | -2.3 (2.12)
  Day 14, n=61 | -2.2 (2.21)
  Day 15, n=61 | -2.5 (2.12)
  Day 16, n=61 | -2.3 (2.05)
  Day 17, n=61 | -2.4 (2.01)
  Day 18, n=61 | -2.5 (1.96)
  Day 19, n=61 | -2.6 (2.01)
  Day 20, n=61 | -2.7 (2.00)
  Day 21, n=61 | -2.5 (2.08)
  Day 22, n=61 | -2.6 (2.03)
  Day 23, n=61 | -2.4 (2.04)
  Day 24, n=61 | -2.4 (2.13)
  Day 25, n=61 | -2.5 (1.91)
  Day 26, n=61 | -2.5 (2.08)
  Day 27, n=61 | -2.5 (1.97)
  Day 28, n=61 | -2.4 (1.99)
  Day 29, n=60 | -2.4 (1.81)
  Day 30, n=60 | -2.5 (1.79)
  Day 31, n=60 | -2.6 (1.90)
  Day 32, n=60 | -2.4 (2.16)
  Day 33, n=60 | -2.5 (1.99)
  Day 34, n=60 | -2.4 (2.30)
  Day 35, n=60 | -2.4 (2.43)
  Day 36, n=60 | -2.2 (2.21)
  Day 37, n=60 | -2.4 (2.23)
  Day 38, n=60 | -2.4 (2.41)
  Day 39, n=60 | -2.2 (2.30)
  Day 40, n=60 | -2.2 (2.17)
  Day 41, n=60 | -2.3 (1.85)
  Day 42, n=60 | -2.6 (1.80)
  Day 43, n=60 | -2.4 (2.20)
  Day 44, n=60 | -2.5 (2.16)
  Day 45, n=60 | -2.2 (2.24)
  Day 46, n=60 | -2.5 (1.89)
  Day 47, n=60 | -2.5 (2.07)
  Day 48, n=60 | -2.4 (2.27)
  Day 49, n=60 | -2.4 (2.15)
  Day 50, n=60 | -2.4 (2.33)
  Day 51, n=60 | -2.4 (2.34)
  Day 52, n=60 | -2.4 (1.99)
  Day 53, n=60 | -2.5 (1.90)
  Day 54, n=60 | -2.2 (1.98)
  Day 55, n=60 | -2.2 (2.11)
  Day 56, n=60 | -2.3 (2.11)
  Day 57, n=60 | -2.4 (1.94)
  Day 58, n=60 | -2.4 (1.98)
  Day 59, n=60 | -2.6 (2.09)
  Day 60, n=60 | -2.8 (1.75)
  Day 61, n=60 | -2.5 (1.78)
  Day 62, n=60 | -2.6 (1.65)
  Day 63, n=60 | -2.7 (1.77)
  Day 64, n=60 | -2.6 (1.96)
  Day 65, n=60 | -2.5 (2.07)
  Day 66, n=60 | -2.2 (2.24)
  Day 67, n=60 | -2.4 (2.10)
  Day 68, n=60 | -2.3 (2.23)
  Day 69, n=60 | -2.4 (1.96)
  Day 70, n=60 | -2.5 (1.79)
  Day 71, n=60 | -2.4 (1.99)
  Day 72, n=60 | -2.1 (1.97)
  Day 73, n=60 | -2.0 (2.17)
  Day 74, n=59 | -1.6 (2.37)
  Day 75, n=59 | -1.8 (2.34)
  Day 76, n=59 | -1.8 (2.56)
  Day 77, n=59 | -2.1 (2.59)
  Day 78, n=59 | -2.1 (2.49)
  Day 79, n=59 | -1.9 (2.35)
  Day 80, n=59 | -1.8 (2.15)
  Day 81, n=50 | -1.9 (2.25)
  Day 82, n=43 | -1.7 (2.45)
  Day 83, n=39 | -1.2 (2.55)
  Day 84, n=31 | -1.2 (2.55)

14. Secondary Outcome: Mean Change From Baseline in the 4 Total Nasal Symptom Score (4TNSS) Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: The 4TNSS is the sum of the 4 individual symptom scores for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is scored on a scale from 0 to 3; the range of sums for the 4TNSS is 0 to 12. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average of the 4TNSS in the last 4 consecutive days prior to Visit 2 (start of the treatment period). A mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Scores on a scale | -2.6 (2.01)
  Week 1 to 2 n=61 | -1.8 (1.93)
  Week 3 to 4, n=61 | -2.9 (2.26)
  Week 7 to 8, n=60 | -2.8 (2.26)
  Week 11 to 12, n=60 | -2.3 (2.50)

15. Secondary Outcome: Mean Percent Change From Baseline in the 4 Total Nasal Symptom Score (4TNSS) Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: The 4TNSS is the sum of the 4 individual symptom scores for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is scored on a scale from 0 to 3; the range of sums for the 4TNSS is 0 to 12. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average of the 4TNSS in the last 4 consecutive days prior to Visit 2 (start of the treatment period). A mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from Baseline=(mean score at the post-Baseline assessment minus the score at Baseline) divided by the Baseline value * 100.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Percent change
  Entire Treatment Period, n=61 | -47.1 (34.06)
  Week 1 to 2, n=61 | -31.3 (38.42)
  Week 3 to 4, n=61 | -52.8 (38.62)
  Week 7 to 8, n=60 | -51.3 (38.90)
  Week 11 to 12, n=60 | -42.0 (41.95)

16. Secondary Outcome: Mean Change From Baseline in the Total Ocular Symptom Score (TOSS) Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: Symptoms of eye itching, tearing, and redness were scored by the participant's parent/guardian who signed the ICF or the participant themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the participant's diary. The TOSS is the sum of all three symtpom scores and ranges from 0 to 9. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Entire Treatment Period, n=61 | -0.2 (1.00)
  Week 1 to 2, n=61 | -0.1 (0.88)
  Week 3 to 4, n=61 | -0.1 (1.08)
  Week 7 to 8, n=60 | -0.2 (1.20)
  Week 11 to 12, n=60 | -0.3 (1.06)

17. Secondary Outcome: Mean Percent Change From Baseline in the Total Ocular Symptom Score (TOSS) Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: Symptoms of eye itching, tearing, and redness were scored by the participant's parent/guardian who signed the ICF or the participant themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the participant's diary. The TOSS is the sum of all three symtpom scores and ranges from 0 to 9. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from Baseline=(mean score at the post-Baseline assessment minus the score at Baseline) divided by the Baseline value * 100.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Percent change
  Entire Treatment Period, n=36 | 7.1 (180.60)
  Week 1 to 2, n=36 | 4.6 (138.41)
  Week 3 to 4, n=36 | 17.5 (214.79)
  Week 7 to 8, n=35 | 29.0 (251.46)
  Week 11 to 12, n=35 | -22.5 (163.35)

18. Secondary Outcome: Mean Change From Baseline in Sneezing, Rhinorrhea, Nasal Congestion, and Nasal Itching Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: Four individual symptoms (sneezing, rhinorrhea, nasal congestion, and nasal itching) were scored on a scale from 0 to 3 using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average of the symptom scores in the last 4 consecutive days prior to Visit 2 (start of the treatment period). A mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Sneezing, Entire Treatment Period, n=61 | -0.7 (0.74)
  Sneezing, Week 1 to 2, n=61 | -0.5 (0.67)
  Sneezing, Week 3 to 4, n=61 | -0.8 (0.75)
  Sneezing, Week 7 to 8, n=60 | -0.7 (0.81)
  Sneezing, Week 11 to 12, n=60 | -0.6 (0.88)
  Rhinorrhea, Entire Treatment Period, n=61 | -0.8 (0.65)
  Rhinorrhea, Week 1 to 2, n=61 | -0.5 (0.62)
  Rhinorrhea, Week 3 to 4, n=61 | -0.9 (0.76)
  Rhinorrhea, Week 7 to 8, n=60 | -0.8 (0.73)
  Rhinorrhea, Week 11 to 12, n=60 | -0.7 (0.85)
  Nasal Congestion, Entire Treatment Period, n=61 | -0.8 (0.66)
  Nasal Congestion, Week 1 to 2, n=61 | -0.5 (0.63)
  Nasal Congestion, Week 3 to 4, n=61 | -0.9 (0.76)
  Nasal Congestion, Week 7 to 8, n=60 | -0.8 (0.72)
  Nasal Congestion, Week 11 to 12, n=60 | -0.7 (0.85)
  Nasal Itching, Entire Treatment Period, n=61 | -0.4 (0.58)
  Nasal Itching, Week 1 to 2, n=61 | -0.2 (0.55)
  Nasal Itching, Week 3 to 4, n=61 | -0.4 (0.63)
  Nasal Itching, Week 7 to 8, n=60 | -0.4 (0.67)
  Nasal Itching, Week 11 to 12, n=60 | -0.3 (0.69)

19. Secondary Outcome: Mean Change From Baseline in Eye Itching, Tearing, and Redness Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: Three individual symptoms (eye itching, tearing, and redness) were scored by the participant's parent/guardian who signed the ICF or the participant themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the participant's diary. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Eye Itching, Entire Treatment Period, n=61 | -0.2 (0.57)
  Eye Itching, Week 1 to 2, n=61 | -0.1 (0.53)
  Eye Itching, Week 3 to 4, n=61 | -0.1 (0.61)
  Eye Itching, Week 7 to 8, n=60 | -0.2 (0.68)
  Eye Itching, Week 11 to 12, n=60 | -0.2 (0.59)
  Tearing, Entire Treatment Period, n=61 | 0.0 (0.25)
  Tearing, Week 1 to 2, n=61 | 0.0 (0.22)
  Tearing, Week 3 to 4, n=61 | 0.0 (0.29)
  Tearing, Week 7 to 8, n=60 | 0.0 (0.28)
  Tearing, Week 11 to 12, n=60 | 0.0 (0.26)
  Redness, Entire Treatment Period, n=61 | -0.1 (0.34)
  Redness, Week 1 to 2, n=61 | -0.0 (0.32)
  Redness, Week 3 to 4, n=61 | -0.0 (0.35)
  Redness, Week 7 to 8, n=60 | -0.0 (0.43)
  Redness, Week 11 to 12, n=60 | -0.1 (0.39)

20. Secondary Outcome: Mean Change From Baseline in the Score of Troubles With Daily Life Over the Entire Treatment Period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Description: The participant's parent/guardian who signed the ICF or the participant themself scored the participant's troubles with daily life once daily using the following scale: 0, None; 1, Few troubles; 2, Intermediate between 3 and 1; or 3, Painful and complicating daily life. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period, Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (12 weeks), Week 1 to 2, Week 3 to 4, Week 7 to 8, and Week 11 to 12
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
Scores on a scale
  Entire Treatment Period, n=61 | -0.5 (0.61)
  Week 1 to 2, n=61 | -0.3 (0.52)
  Week 3 to 4, n=61 | -0.5 (0.65)
  Week 7 to 8, n=60 | -0.6 (0.72)
  Week 11 to 12, n=60 | -0.4 (0.75)

21. Secondary Outcome: Number of Participants With the Indicated Scores for Rhinoscopy Findings (Swelling of Inferior Turbinate Mucosa, Color of Inferior Turbinate Mucosa, Quantity of Nasal Discharge, and Quality of Nasal Discharge)
Description: Rhinoscopy was assessed by the investigator by scoring swelling of inferior turbinate mucosa (SOITM) scored as 0 (none), 1 (possible to see center of the middle turbinate), 2 (between 3 and 1), or 3 (impossible to see middle turbinate); color of inferior turbinate mucosa (COITM) scored as 0 (normal), 1 (pink), 2 (red), or 3 (pale); quantity of nasal discharge (QTND) scored as 0 (none), 1 (small amount adhered), 2 (between 3 and 1), or 3 (filled); and quality of nasal discharge (QLND) scored as 0 (none), 1 (pyoid), 2 (viscous), or 3 (watery).
Time Frame: Baseline, Week 4, Week 8, and Week 12/early withdrawal
Population: FAS Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: participants
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
participants
  SOITM, Baseline, Score 0, n=61 | 3
  SOITM, Baseline, Score 1, n=61 | 9
  SOITM, Baseline, Score 2, n=61 | 35
  SOITM, Baseline, Score 3, n=61 | 14
  SOITM, Week 4, Score 0, n=60 | 15
  SOITM, Week 4, Score 1, n=60 | 21
  SOITM, Week 4, Score 2, n=60 | 23
  SOITM, Week 4, Score 3, n=60 | 1
  SOITM, Week 8, Score 0, n=60 | 17
  SOITM, Week 8, Score 1, n=60 | 24
  SOITM, Week 8, Score 2, n=60 | 19
  SOITM, Week 8, Score 3, n=60 | 0
  SOITM, Week 12/early withdrawal, Score 0, n=61 | 21
  SOITM, Week 12/early withdrawal, Score 1, n=61 | 26
  SOITM, Week 12/early withdrawal, Score 2, n=61 | 13
  SOITM, Week 12/early withdrawal, Score 3, n=61 | 1
  COITM, Baseline, Score 0, n=61 | 0
  COITM, Baseline, Score 1, n=61 | 10
  COITM, Baseline, Score 2, n=61 | 23
  COITM, Baseline, Score 3, n=61 | 28
  COITM, Week 4, Score 0, n=60 | 10
  COITM, Week 4, Score 1, n=60 | 28
  COITM, Week 4, Score 2, n=60 | 13
  COITM, Week 4, Score 3, n=60 | 9
  COITM, Week 8, Score 0, n=60 | 12
  COITM, Week 8, Score 1, n=60 | 30
  COITM, Week 8, Score 2, n=60 | 11
  COITM, Week 8, Score 3, n=60 | 7
  COITM, Week 12/early withdrawal, Score 0, n=61 | 19
  COITM, Week 12/early withdrawal, Score 1, n=61 | 28
  COITM, Week 12/early withdrawal, Score 2, n=61 | 10
  COITM, Week 12/early withdrawal, Score 3, n=61 | 4
  QTND, Baseline, Score 0, n=61 | 4
  QTND, Baseline, Score 1, n=61 | 16
  QTND, Baseline, Score 2, n=61 | 33
  QTND, Baseline, Score 3, n=61 | 8
  QTND, Week 4, Score 0, n=60 | 30
  QTND, Week 4, Score 1, n=60 | 24
  QTND, Week 4, Score 2, n=60 | 5
  QTND, Week 4, Score 3, n=60 | 1
  QTND, Week 8, Score 0, n=60 | 29
  QTND, Week 8, Score 1, n=60 | 25
  QTND, Week 8, Score 2, n=60 | 4
  QTND, Week 8, Score 3, n=60 | 2
  QTND, Week 12/early withdrawal, Score 0, n=61 | 34
  QTND, Week 12/early withdrawal, Score 1, n=61 | 24
  QTND, Week 12/early withdrawal, Score 2, n=61 | 3
  QTND, Week 12/early withdrawal, Score 3, n=61 | 0
  QLND, Baseline, Score 0, n=61 | 4
  QLND, Baseline, Score 1, n=61 | 0
  QLND, Baseline, Score 2, n=61 | 14
  QLND, Baseline, Score 3, n=61 | 43
  QLND, Week 4, Score 0, n=60 | 30
  QLND, Week 4, Score 1, n=60 | 11
  QLND, Week 4, Score 2, n=60 | 4
  QLND, Week 4, Score 3, n=60 | 15
  QLND, Week 8, Score 0, n=60 | 30
  QLND, Week 8, Score 1, n=60 | 13
  QLND, Week 8, Score 2, n=60 | 5
  QLND, Week 8, Score 3, n=60 | 12
  QLND, Week 12/early withdrawal, Score 0, n=61 | 32
  QLND, Week 12/early withdrawal, Score 1, n=61 | 10
  QLND, Week 12/early withdrawal, Score 2, n=61 | 7
  QLND, Week 12/early withdrawal, Score 3, n=61 | 12

22. Secondary Outcome: Number of Participants With the Indicated Overall Response to Therapy, as Assessed by the Investigator
Description: The investigator evaluated the participant's overall response to therapy (defined as improvement in the symptoms of allergic rhinitis) compared with Visit 2 (start of the treatment period), using the following 7-point categorical scale: 1=significantly improved, 2=moderately improved, 3=mildly improved, 4=no change, 5=mildly worse, 6=moderately worse, and 7=significantly worse.
Time Frame: Week 12/early withdrawal
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
participants
  Significantly Improved | 25
  Moderately Improved | 28
  Mildly Improved | 3
  No Change | 5
  Mildly Worse | 0
  Moderately Worse | 0
  Significantly Worse | 0

23. Secondary Outcome: Number of Participants With the Indicated Overall Response to Therapy, as Assessed by the Participant's Parent/Guardian or the Participant
Description: The participant's parent/guardian who signed the ICF or the participant himself/herself evaluated the participant's overall response to therapy (defined as improvement in the symptoms of allergic rhinitis) compared with Visit 2 (start of the treatment period), using the following 7-point categorical scale: 1=significantly improved, 2=moderately improved, 3=mildly improved, 4=no change, 5=mildly worse, 6=moderately worse, and 7=significantly worse.
Time Frame: Week 12/early withdrawal
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 61
participants
  Significantly Improved | 13
  Moderately Improved | 31
  Mildly Improved | 12
  No Change | 4
  Mildly Worse | 1
  Moderately Worse | 0
  Significantly Worse | 0

24. Secondary Outcome: Number of Participants With the Indicated Plasma Concentration of GW685698X for Participants Aged >=2 to <6 Years
Description: Pharmacokinetic (PK) samples were collected to analyze the plasma concentration of GW685698X.
Time Frame: Between 0.5 to 2 hours after final dosing at Week 12 (Visit 5)
Population: PK Concentration Population: all participants from whom a PK sample was obtained and analyzed. Only those participants aged >=2 to <6 years were assessed.
Measure: Number; unit: participants
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 19
participants
  Not Quantifiable (<10 picograms/milliliter [pg/mL] | 17
  >=10 to <20 pg/mL | 2
  >=20 to <30 pg/mL | 0
  >=30 pg/mL | 0

25. Secondary Outcome: Number of Participants With the Indicated Plasma Concentration of GW685698X for Participants Aged >=6 to <15 Years
Description: PK samples were collected to analyze the plasma concentration of GW685698X.
Time Frame: Between 0.5 to 2 hours after final dosing at Week 12 (Visit 5)
Population: PK Concentration Population. Only those participants aged >=6 to <15 years were assessed.
Measure: Number; unit: participants
Arm/Group | GW685698X 55 μg QD
Number analyzed (Participants) | 40
participants
  Not Quantifiable (<10 pg/mL) | 37
  >=10 to <20 pg/mL | 2
  >=20 to <30 pg/mL | 1
  >=30 pg/mL | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment (Visit 2) until follow-up contact (Visit 6) (up to 13 weeks).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of study medication, according to the actual treatment received.
Arm/Group | GW685698X 55 μg QD
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 23/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW685698X 55 μg QD (N=61)
Nasopharyngitis (Infections and infestations) | 15
Acute sinusitis (Infections and infestations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.